CLINICAL TRIAL: NCT01634425
Title: Providing Rapid Out of Hospital Acute Cardiovascular Treatment (PROACT) Novel Proximal Pathways for Non ST Elevation Myocardial Infarction
Brief Title: Providing Rapid Out of Hospital Acute Cardiovascular Treatment (PROACT)
Acronym: PROACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian VIGOUR Centre (Other)
Responsible Party: Principal Investigator, Robert Welsh, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PROACT NSTEMI
Record Dates: First submitted 2011-10-03; First posted 2012-07-06 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: NSTEMI
Keywords: NSTEMI; Point of Care Biomarkers
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - no pre-hospital biomarkers (No Intervention): Standard of Care
- Group 2 - pre-hospital biomarkers (Experimental): Troponin and BNP measured on a POC meter in the ambulance on the way to the hospital.
  Interventions: Device: Alere Triage Meter Pro

INTERVENTIONS:
Device: Alere Triage Meter Pro — Troponin and BNP measured on point of care meter.
  Other Names: Point of Care Meter
  Arms: Group 2 - pre-hospital biomarkers

SUMMARY:
The purpose of this study is to determine if early diagnosis and risk stratification acquired through pre-hospital clinical assessment, 12-lead electrocardiogram and point of care biomarkers will facilitate enhanced triage and treatment in patients with presumed non-ST elevation acute coronary syndromes (NSTEMI).

DETAILED DESCRIPTION:
Utilizing the platform of pre-hospital STEMI research and clinical experience developed over the past decade; we now intend to investigate how best to achieve timely diagnosis and risk stratification of patients that present to pre-hospital emergency medical services with symptoms suspicious for acute NSTEMI through utilization of systematic clinical assessment, pre-hospital 12 lead electrocardiogram and point of care measurement of biomarkers. Additionally, where deemed appropriate these patients will be enrolled in a clinical Chest Pain Protocol utilizing the pre-hospital biomarkers. We hypothesize that establishing a pre-hospital diagnosis in this condition may facilitate efficient triage and -as appropriate- in-hospital disposition. Additionally, the enhanced pre-hospital assessment of this population will facilitate appropriate timely disposition of those patients not found to have acute cardiovascular disease. These processes will facilitate decanting the frequently overcrowded and under resources Emergency Departments.

ELIGIBILITY:
Inclusion Criteria

1. Patient that activates pre-hospital Emergency Medical Services (EMS) for symptoms of acute chest discomfort for which acute cardiovascular disease is deemed to be the most probable diagnosis by EMS personnel.
2. Patient is older than 30 years of age
3. Patient is able to give informed consent

Exclusion Criteria

1. Patient with documented ST elevation on the initial 12 lead ECG
2. Patient with a prior diagnosis that is compatible with another disease i.e. severe asthma, etc.
3. Patient with Central Nervous System symptoms or syncope
4. Patient with cardiac arrest, ventricular tachycardia or atrial fibrillation with heart rate > 110 bpm

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2011-11; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Time from first medical contact to final patient disposition. | From date of first medical contact until first appropriate therapy given, assessed up to 30 months
  An Adjudication Committee will examine the records to determine final diagnosis.
  Final patient disposition is defined as the time when a plan for patient discharge from the ED or admission to hospital is both established and documented.

SECONDARY OUTCOMES:
Time to administration of appropriate evidence based therapy | Assessed up to 30 months.
  From time of first medical contact to First appropriate therapy for NSTEMI is defined as: receiving oral antiplatelet agent (excluding ASA - which is routinely administered prior to diagnosis) or intravenous/subcutaneous antithrombotic agents (low molecular weight heparin or IV heparin or glycoprotein IIb/IIIa receptor inhibitors).
Length of hospital stay for patients admitted to hospital | Assessed up to 30 months
In-hospital clinical events (day 7 or discharge) all-cause mortality, cardiogenic shock, heart failure, re-Myocardial infarction | Assessed up to 30 months
30-day all-cause mortality | Assessed up to 30 months
30 day all-cause hospitalization or re-hospitalization | Assessed up to 30 months
30-day composite (all-cause mortality or all-cause hospitalization) | Assessed up to 30 months

OTHER OUTCOMES:
Explore the incremental value pre-hospital BNP on primary and secondary endpoints. | Assessed up to 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Armstrong, MD, Study Chair — Canadian VIGOUR Centre
Locations (5):
- Canada (5):
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Northeast Community Health Centre (NECHC), Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta

REFERENCES:
- [Derived] Sepehrvand N, Zheng Y, Armstrong PW, Welsh RC, Ezekowitz JA. Identifying Low-risk Patients for Early Discharge From Emergency Department Without Using Subjective Descriptions of Chest Pain: Insights From Providing Rapid Out of Hospital Acute Cardiovascular Treatment (PROACT) 3 and 4 Trials. Acad Emerg Med. 2017 Jun;24(6):691-700. doi: 10.1111/acem.13183. Epub 2017 May 12. PMID 28261896
- [Derived] Ezekowitz JA, Welsh RC, Weiss D, Chan M, Keeble W, Khadour F, Sharma S, Tymchak W, Sookram S, Brass N, Knapp D, Koshy TL, Zheng Y, Armstrong PW. Providing Rapid Out of Hospital Acute Cardiovascular Treatment 4 (PROACT-4). J Am Heart Assoc. 2015 Dec 1;4(12):e002859. doi: 10.1161/JAHA.115.002859. PMID 26627881
- [Derived] Sepehrvand N, Zheng Y, Armstrong PW, Welsh R, Goodman SG, Tymchak W, Khadour F, Chan M, Weiss D, Ezekowitz JA. Alignment of site versus adjudication committee-based diagnosis with patient outcomes: Insights from the Providing Rapid Out of Hospital Acute Cardiovascular Treatment 3 trial. Clin Trials. 2016 Apr;13(2):140-8. doi: 10.1177/1740774515601437. Epub 2015 Aug 19. PMID 26289822